CLINICAL TRIAL: NCT01798342
Title: Gastric Residual Volume After He Intake Of Maltodextrin And Glutamine. A Randomized Double-Blind, Crossover Study
Brief Title: Safety of Gastric Volume Emptying After the Intake of Maltodextrin and Glutamine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of Mato Grosso (Other)
Responsible Party: Principal Investigator, Jose Eduardo de Aguilar-Nascimento, Professor, Federal University of Mato Grosso
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: brianez
Record Dates: First submitted 2013-02-19; First posted 2013-02-25 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Pulmonary Aspiration of Gastric Contents; Adverse Effects in the Therapeutic Use of Other and Unspecified General Anaesthetics; Pulmonary Aspiration During Anaesthetic Induction
Keywords: preoperative care; maltodextrine; glutamine; gastric residual volume; MRI
MeSH Terms: conditions — Respiratory Aspiration of Gastric Contents | interventions — maltodextrin; Glutamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Maltodextrin (Active Comparator): The volunteers ingested 400ml (4 hours before the exam was carried out) at 8:00AM and 200ml (2 hours before the exam was carried out) at 10:00AM of a beverage containing water plus 12.5% maltodextrin
  Interventions: Dietary Supplement: Maltodextrin
- Glutamine (Experimental): The same volunteers ingested 400ml (4 hours before the exam was carried out) at 8:00AM and 200ml (2 hours before the exam was carried out) at 10:00AM of a beverage containing water plus 12.5% maltodextrin plus 15g of glutamine
  Interventions: Dietary Supplement: Glutamine

INTERVENTIONS:
Dietary Supplement: Maltodextrin — The volunteers underwent MRI after the ingestion of the dietary supplement in a crossover fashion aiming at measuring the gastric residual volume
  Other Names: Maltodestrin plus glutamine
  Arms: Maltodextrin
Dietary Supplement: Glutamine — The volunteers ingested 400ml (4 hours before the exam was carried out) at 8:00AM and 200ml (2 hours before the exam was carried out) at 10:00AM of a beverage containing water plus 12.5% maltodextrin plus 15g of GLN before MRI
  Arms: Glutamine

SUMMARY:
Carbohydrates (CHO)-based drinks 2h before the induction of anesthesia are recommended to decrease insulin resistance. The addition of glutamine (GLN) in these beverages may enhance the benefits of CHO alone. However, only a few studies tested the safety of this formula. The objective of this study was to evaluate the gastric residual volume (GRV) after the intake of a beverage containing CHO plus GLN using magnetic resonance (MRI).

DETAILED DESCRIPTION:
We included 11 male young volunteers (aged between 21 and 30 years-old) with body mass index (BMI) between 20 and 29 kg/m2 and without either acute or chronic illness in the last 3 months. The criteria for exclusion were non-adherence to any phase of the study protocol, gastroesophageal reflux disease, previous history of intolerance to lactose, gastroparesis or history of poor gastric emptying, diabetes mellitus, and previous abdominal surgery.

Each volunteer was randomized for participation in the study in a blind fashion. All subjects underwent two different protocols before MRI with an interval of seven days between them. Both phases took place after an overnight fast of eight hours. The volunteers ingested 400ml (4 hours before the exam was carried out) at 8:00AM and 200ml (2 hours before the exam was carried out) at 10:00AM of a beverage containing either water plus 12.5% maltodextrin (Phloraceae, Cuiabá, Brazil; CHO group) or the same beverage plus 15g of GLN (Phloraceae, Cuiabá, Brazil; GLN group). The participants were instructed not to ingest alcohol, medication, and caffeine within 24 hours of the study, nor do any vigorous physical activity during that time.

In both phases the individuals were blind to the specific drink and they were told to ingest the beverage in a maximum period of five minutes and T0 was defined as the moment they complete the intake of the solution.The powdered products (maltodextrin alone or maltodextrine plus glutamine) were packed in coded opaque sachets and the content was only known by the pharmacist who manipulated it.

All the participants in the study underwent magnetic resonance of the upper abdomen at 12:00AM and 01:00PM. The GRV observed during the first exam was defined as T120 and the second exam as T180. All exams were performed by the same magnetic resonance equipment (Intera 1.5T ; Philips Healthcare, Eindhoven, Holland).

ELIGIBILITY:
Inclusion Criteria:

* Young male volunteers (aged between 21 and 30 years-old) with body mass index (BMI) between 20 and 29 kg/m2 and without either acute or chronic illness in the last 3 months.

Exclusion Criteria:

* non-adherence to any phase of the study protocol,
* gastroesophageal reflux disease,
* previous history of intolerance to lactose,
* gastroparesis or history of poor gastric emptying,
* diabetes mellitus, and
* previous abdominal surgery

Ages: 21 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2012-03; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Gastric residual volume (GVR) ("change" is being assessed) | immediately after ingestion (T0), 120 minutes after (T120) and 180 (T180) minutes after ingestion
  We measured the GRV by MRI immediately after ingestion (T0)and the changes of GVR after 120 (T120)and 180 minutes (T180)- "change" is being assessed

SECONDARY OUTCOMES:
Vomiting | 180 minutes
  We observed whether the volunteer presented vomiting during the experiment

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Santa Rosa, Cuiabá, Mato Grosso, Brazil